CLINICAL TRIAL: NCT03973814
Title: Hypothermia Risk With Continuous Renal Replacement Therapy
Acronym: HR-CRRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Max Bell, MD, PhD, Principal Investigator, Karolinska University Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: BxIIRgrant
Record Dates: First submitted 2019-05-30; First posted 2019-06-04 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Acute Kidney Injury; Hypothermia
Keywords: continuous renal replacement therapy
MeSH Terms: conditions — Acute Kidney Injury; Hypothermia

STUDY DESIGN:
Intervention Model Description: The investigators will assess body temperature before-, during- and after Thermax blood warming treatment. Patients are essentially their own controls.
  Moreover, we will use historic data on the previous blood warmer for the Prismaflex device to assess temperature changes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Prior to Thermax Warming (Active Comparator): Baseline temperature
  Interventions: Device: Thermax Blood Warmer
- During warming (Active Comparator): Temperature during Thermax warming
  Interventions: Device: Thermax Blood Warmer
- Post warming (Active Comparator): Temperature after cessation of Thermax warming
  Interventions: Device: Thermax Blood Warmer

INTERVENTIONS:
Device: Thermax Blood Warmer — Patients will be their own controls: Prior to-, during-, and after Thermax blood warming.

SUMMARY:
The present study aims at testing if the TherMax blood warmer is more accurate and reliable in reaching and maintaining chosen target temperature during continuous renal replacement therapy as compared to the Prismaflo IIS blood warmer used for the PrismaFlex system.

DETAILED DESCRIPTION:
Blood warming devices during continuous renal replacement therapy (CRRT) have not been adequately tested.

The novel TherMax blood warmer for the newly introduced PrisMax System heats blood and replacement solutions via a dry heat plate system. In contrast, the PRISMAFLO IIS Blood Warmer for PRISMAFLEX System uses an electric heating sleeve on a standard CRRT filter set.

Data on adverse events (AE) during continuous renal replacement therapy (CRRT) has been studied and one of the most common AE was hypothermia, reported in 44% of all cases.

The present study aims at testing if the TherMax blood warmer is more accurate and reliable in reaching and maintaining chosen target temperature during CRRT as compared to the blood warmer used for the PrismaFlex system.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-100 years) critically ill patients treated with CRRT.

Exclusion Criteria:

* Patients under 18 years of age. Non-RRT patients.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Temperature, accuracy | 24 hours
  During use of Thermax; hourly difference between prescribed temperature-measured temperature; accuracy 0,1 Celsius

SECONDARY OUTCOMES:
Temperature, differences | 12-18 hours (six hour warming period)
  Difference to 36.5 Celsius, std deviation, interquartile range: Prior to Thermax, during Thermax and after Thermax
Historic comparator | 24 hours
  Using registry/PDMS data, how did the old blood warmer perform with regards to temperature

CONTACTS AND LOCATIONS:
Overall Officials: Max Bell, MD, PhD, Principal Investigator — Karolinska University Hospital; Marcus Broman, MD, PhD, Principal Investigator — Skane University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient and machine data may be made available after study completion, but this depends on the patent holder.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Six months after study completion
Access Criteria: Data access will be reviewed by the PI:s and research group.